CLINICAL TRIAL: NCT02814331
Title: Electrohaemodynamic Activity in Epileptic Children: Combined Video-EEG and Near-infrared Spectroscopy (NIRS) Analysis
Brief Title: Electrohaemodynamic Activity in Epileptic Children : Combined Video-EEG and Near-infrared Spectroscopy (NIRS) Analysis
Acronym: NIRS Epilepsie
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PHRCN11-DR-WALLOIS
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: Video-EEG; near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- symptomatic partial epilepsy: whose brain MRI is abnormal multimodal high-resolution EEG-NIRS
  Interventions: Device: multimodal high-resolution EEG-NIRS
- not symptomatic partial epilepsy: whose brain MRI is normal multimodal high-resolution EEG-NIRS
  Interventions: Device: multimodal high-resolution EEG-NIRS

INTERVENTIONS:
Device: multimodal high-resolution EEG-NIRS

SUMMARY:
Evaluate the contribution of multimodal high-resolution EEG-NIRS electrical and local haemodynamic analysis to spatial localization of epileptogenic foci

DETAILED DESCRIPTION:
This study is designed to evaluate the contribution of multimodal high-resolution EEG-NIRS electrical and local haemodynamic analysis (HR-EEG, HR-NIRS) to spatial localization of epileptogenic foci in order to perform multimodal mapping and localization of interictal spikes (by HR-EEG source reconstruction) with the clinical prospects of guiding the SEEG electrode implantation strategy prior to surgery in children with drug-refractory partial epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 and 18 years
* with drug-refractory partial epilepsy, presenting interictal spikes on standard EEG recordings.

Exclusion Criteria:

* Children with a serious congenital malformation.
* Refusal from one of the parents or the child.
* Children with generalized epilepsy or diffuse interictal spikes.
* Children with severely impaired general status and vital functions.
* Children with dermatosis of the face or scalp.
* Children under the age of 6 years or adults over the age of 18 years.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 6 and 18 years with drug-refractory partial epilepsy, presenting interictal spikes on standard EEG recordings.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-10-14 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
multimodal high-resolution EEG-NIRS | Day 0
  to evaluate the contribution of multimodal high-resolution EEG-NIRS electrical and local haemodynamic analysis (HR-EEG, HR-NIRS) to spatial localization of epileptogenic foci in order to perform multimodal mapping and localization of interictal spikes (by HR-EEG source reconstruction) with the clinical prospects of guiding the SEEG electrode implantation strategy prior to surgery in children with drug-refractory partial epilepsy.

SECONDARY OUTCOMES:
Functional MRI | Day 0
  to analyse the temporal dynamics of haemodynamic changes surrounding epileptic spikes.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice WALLOIS, Md, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France